CLINICAL TRIAL: NCT02158312
Title: Bihemispheric Modulation of the Motor Cortex by Single-session Transcranial Direct Current Stimulation During Training in Subacute Stroke Patients
Brief Title: Bihemispheric Modulation of the Motor Cortex by Transcranial Direct Current Stimulation in Subacute Stroke Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2014-01-006C
Record Dates: First submitted 2014-06-04; First posted 2014-06-06 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-06

CONDITIONS: Stroke
Keywords: neuroplasticity
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- transcranial direct current stimulation (Experimental): bihemispheric transcranial direct current stimulation, anodal at ipsilesional M1 while cathodal at contralesional M1, for 20 minutes
  Interventions: Device: Magstim Eldith DC-stimulator(Magstim Co., Whitland, UK)
- sham stimulation (Placebo Comparator): same as the experimental stimulation condition but only for 2 minutes

INTERVENTIONS:
Device: Magstim Eldith DC-stimulator(Magstim Co., Whitland, UK) — 2 mA for 20 minutes transcranial direct current stimulation
  Arms: transcranial direct current stimulation

SUMMARY:
Post-stroke sensorimotor recovery largely depends on ipsilesional and interhemispheric motor circuit reorganization. Transcranial direct current stimulation (tDCS) may be used to enhance after-effects of rehabilitation through membrane polarization modulation. In this double-blind, crossover randomized controlled trial, we aim to investigate whether single-session, bihemispheric tDCS to the primary motor cortex (M1) in combination with upper extremity rehabilitation therapy modulates ipsilesional motor circuit excitability using transcranial magnetic stimulation (TMS) and magnetoencephalography (MEG) measures.

DETAILED DESCRIPTION:
We will consecutively enroll subacute (2-4 weeks after stroke onset) patients with first-time, unilateral, ischemic subcortical stroke in the middle cerebral artery territory with mild to moderate hand weakness. All subjects will be assessed for baseline upper extremity motor function (Fugl-Meyer test and Action Research Arm test), structural and functional magnetic resonance imaging (fMRI). A single session of bihemispheric tDCS (anodal tDCS to ipsilesional M1 and cathodal tDCS to contralesional M1 with 2 mA stimulation for 20 min) or sham tDCS (same but stimulation for only 2 min) with simultaneous physical/occupational therapy will be tested in each subject with a randomized sequence on different days (at least two days apart from each other). All stroke patients will receive standard medical and rehabilitation treatments during the study period. Changes in corticospinal excitability and transcallosal inhibition from the TMS study, as well as sensorimotor oscillations, MEG source projection, and functional connectivity from the task-related MEG will be assessed immediately before and after intervention.

ELIGIBILITY:
Inclusion Criteria:

* subacute (2-4 weeks after stroke onset) patients
* first-time, unilateral, ischemic subcortical stroke in the middle cerebral artery territory
* mild to moderate hand weakness (MRC 2-4/5)

Exclusion Criteria:

* cerebral cortex lesions
* containing metal implants (such as implanted electrodes, pacemakers)
* sensitive or fear of electromagnetic waves
* pregnant women
* history of alcohol or drug abuse
* history of seizures or epilepsy EEG recording
* other significant disease or neuropsychiatric disorders
* claustrophobia
* fixed dentures over two or more (enough to interfere with MEG signals)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-05; Primary Completion 2017-05 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
transcranial magnetic stimulation (TMS) | up to 20 minutes

CONTACTS AND LOCATIONS:
Overall Officials: I-Hui Lee, MD PhD, Principal Investigator — Department of Neurology, Taipei Veterans General Hospital, Taipei, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan